CLINICAL TRIAL: NCT03679949
Title: Effects of Cannabis on Prescription Drug Abuse Liability and Analgesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Caroline A. Arout, Ph.D., Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 7647
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Pain; Abuse, Drug
Keywords: experimental pain; Cannabis; Cannabidiol; THC
MeSH Terms: conditions — Pain; Substance-Related Disorders; Marijuana Abuse | interventions — Oxycodone; nabiximols

STUDY DESIGN:
Intervention Model Description: This is a randomized, cross-over, double-blind, placebo-controlled study. All participants will partake in each arm and receive all interventions.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Placebo (Placebo Comparator): Participants will receive 0 mg oxycodone (oral) and placebo cannabis (vaporized)
  Interventions: Drug: Placebo
- Oxycodone (Experimental): Participants will receive 2.5 mg oxycodone (oral) and placebo cannabis (vaporized)
  Interventions: Drug: Oxycodone; Drug: Placebo
- Cannabis (THC:CBD = ~1:0) (Experimental): Participants will receive 0 mg oxycodone (oral) and cannabis with high THC concentrations (vaporized)
  Interventions: Drug: Cannabis (THC:CBD = ~ 1:0); Drug: Placebo
- Cannabis (THC:CBD = ~ 0:1) (Experimental): Participants will receive 0 mg oxycodone (oral) and cannabis with high CBD concentrations (vaporized)
  Interventions: Drug: Cannabis (THC:CBD = ~ 0:1); Drug: Placebo
- Cannabis (THC:CBD = ~ 1:1) (Experimental): Participants will receive 0 mg oxycodone (oral) and cannabis with equal CBD and THC concentrations (vaporized)
  Interventions: Drug: Cannabis (THC:CBD = ~ 1:1); Drug: Placebo
- Cannabis (THC:CBD = ~1:0) + Oxycodone (Experimental): Participants will receive 2.5 mg oxycodone (oral) and cannabis with high THC concentrations (vaporized)
  Interventions: Drug: Oxycodone; Drug: Cannabis (THC:CBD = ~ 1:0)
- Cannabis (THC:CBD = ~ 0:1) + Oxycodone (Experimental): Participants will receive 2.5 mg oxycodone (oral) and cannabis with high CBD concentrations (vaporized)
  Interventions: Drug: Oxycodone; Drug: Cannabis (THC:CBD = ~ 0:1)
- Cannabis (THC:CBD = ~ 1:1) + Oxycodone (Experimental): Participants will receive 2.5 mg oxycodone (oral) and cannabis with equal concentrations of THC and CBD (vaporized)
  Interventions: Drug: Oxycodone; Drug: Cannabis (THC:CBD = ~ 1:1)

INTERVENTIONS:
Drug: Oxycodone — Oxycodone, 2.5 mg
  Arms: Cannabis (THC:CBD = ~ 0:1) + Oxycodone; Cannabis (THC:CBD = ~ 1:1) + Oxycodone; Cannabis (THC:CBD = ~1:0) + Oxycodone; Oxycodone
Drug: Cannabis (THC:CBD = ~ 1:0) — Cannabis with high THC concentration and negligible CBD concentrations
  Arms: Cannabis (THC:CBD = ~1:0); Cannabis (THC:CBD = ~1:0) + Oxycodone
Drug: Cannabis (THC:CBD = ~ 0:1) — Cannabis with high CBD concentration and negligible THC concentrations
  Arms: Cannabis (THC:CBD = ~ 0:1); Cannabis (THC:CBD = ~ 0:1) + Oxycodone
Drug: Cannabis (THC:CBD = ~ 1:1) — Cannabis with equivalent CBD and THC concentrations
  Arms: Cannabis (THC:CBD = ~ 1:1); Cannabis (THC:CBD = ~ 1:1) + Oxycodone
Drug: Placebo — Cannabis with negligible amounts of THC and CBD 0.0 mg oxycodone
  Other Names: Placebo cannabis
  Arms: Cannabis (THC:CBD = ~ 0:1); Cannabis (THC:CBD = ~ 1:1); Cannabis (THC:CBD = ~1:0); Oxycodone; Placebo

SUMMARY:
The purpose of this research is to assess the impact of cannabis on the analgesic and abuse-liability effects of a sub-threshold dose of a commonly used analgesic.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female aged 21-53 years
* Previous cannabis use
* Previous opioid use
* Urine test positive for recent cannabis use
* Being able to perform all study procedures
* Currently practicing an effective form of birth control (women only)

Exclusion Criteria:

* Meeting criteria for some Use Disorders
* Report regular illicit drug use
* If medical history, physical and psychiatric examination, or laboratory tests performed during the screening process revealed any significant illness

Ages: 21 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Subjective Effects | 6 weeks
  Participants will rate "drug liking", "good drug effects", and "high" on a visual analogue scale (VAS; 1-100mm).
Cold Pressor Test | 6 weeks
  Participants will immerse their hand in a bucket of ice water to determine pain threshold and pain tolerance latencies (in seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Caroline A Cooper, PhD, Principal Investigator — New York Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided